CLINICAL TRIAL: NCT07191691
Title: Observational Study of Psychomotor Development in Children Born in France to Parents Born in Sub-Saharan Africa.
Acronym: DEVMOTSUD
Status: Not yet recruiting | Type: Observational
Sponsor: Etablissement Public de Santé Barthélemy Durand (Other)
Responsible Party: Sponsor
Other Study IDs: 22P02; 2025-A00487-42 (Registry Identifier: ANSM)
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Psychomotor Performance; Child Development; Culture
Keywords: Psychomotricity; Child Development; Culture; Migration; Bayley Scales of Infant and toddler Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children born in France to parents born in Sub-Saharan Africa: Subject evaluation included during 60 to 90 minutes. Step 1: The investigator will complete a socio-demographic questionnaire based on the parents' responses.
  Step 2: The BSID-4 (Bayley Scales of Infant and Toddler Development, Fourth Edition) will be completed through observation of the child's behavior. Parents will remain with their child throughout the assessment. The test concludes after five consecutive failures on the final scale administered. Step 3: Subjects will exit the research protocol upon completion of the BSID-4 assessment.
  Interventions: Diagnostic Test: Bayley Scales of Infant and toddler Development, fourth edition (BSID-4)

INTERVENTIONS:
Diagnostic Test: Bayley Scales of Infant and toddler Development, fourth edition (BSID-4) — The BSID-4 is a test that evaluates three areas of child's development, divided into three scales:
  * The Motor Scale, which includes the fine motor and gross motor subtests;
  * The Cognitive Scale, which consists of items assessing sensorimotor development, object exploration and manipulation, concept formation, memory, and other primary functions from which the child's reasoning abilities emerge;
  * The Language Scale, which includes the receptive communication and expressive communication subtests.
  The administration of the BSID-4 involves the standardized delivery of items. The BSID-4 standardization does not specify a fixed order for administering the scales: depending on the child's temperament and spontaneous interest, the examiner adapts the order in which the motor, language, and cognitive scales are administered.

SUMMARY:
The goal of this observational study is to determine whether there are specific characteristics of psychomotor development in children born in France to parents born in Sub-Saharan Africa, using the Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4).

The main question it aims to answer :

Is there a difference in the average raw scores on the motor scale between children born in France to parents from Sub-Saharan Africa and the French standard of the Bayley-4?

Child participants will be included in the study, and their parents will complete a socio-demographic questionnaire. The children will then be observed by the investigator in an enriched environment for 60 to 90 minutes. If necessary, the investigator may provide verbal stimulation.

The children will not be physically manipulated by the investigator, and breaks may be taken at any time as needed. Once the observation is complete, the participant's involvement in the study will end.

DETAILED DESCRIPTION:
Context From the 1950s to the 1970s, studies conducted in Sub-Saharan Africa showed that children acquired independent walking skills at an earlier age. Anthropological research carried out between 1970 and 2000 highlighted differences in mothering practices, shaped by the cultural and environmental context in which children and their parents live.

Since the 2000s, research on child development in Sub-Saharan Africa has increasingly focused on the timing of motor development. The frequency and nature of caregiving practices have been shown to influence the early acquisition of certain skills, while contributing to delays or absence of others. It has therefore been established that the timing and sequence of motor milestones differ between children raised in Sub-Saharan Africa and those raised in France.

In contrast, no data currently exist on the development of children of Sub-Saharan African origin raised in France. Migration-often accompanied by the loss of familiar social and cultural frameworks-is recognized as a significant vulnerability factor. Studies have shown that migration leads to changes in both the frequency and style of caregiving practices.

To date, to the investigators' knowledge, there are no scientific data on the developmental timeline of children born in France to parents from Sub-Saharan Africa (referred to as PNA subjects). However, empirical observations by psychomotor therapists working with PNA children suggest the persistence of certain developmental specificities. One of the most commonly reported signs by parents is early independent walking.

Objectives The primary objective is to determine whether there are specific characteristics of psychomotor development in children born in France to parents born in Sub-Saharan Africa The secondary objective is to establish a timetable of psychomotor development in children born in France to parents born in Sub-Saharan Africa for twenty three items from the developmental early screening standards provided by the government to early childhood professionals.

Hypothesis Is there a difference in the average raw scores on the motor scale between children born in France to parents from Sub-Saharan Africa and the French standard of the Bayley-4?

Methods This study is prospective, comparative, multicenter, non-randomized observational, cohort study

The only visit for included subjects will proceed as follows:

Step 1: The investigator will complete a socio-demographic questionnaire based on the parents' responses.

Step 2: The BSID-4 (Bayley Scales of Infant and Toddler Development, Fourth Edition) will be completed through observation of the child's behavior. Parents will remain with their child throughout the assessment. The test concludes after five consecutive failures on the final scale administered.

Step 3: Subjects will exit the research protocol upon completion of the BSID-4 assessment. The total duration of the single study visit is estimated to be between 60 and 90 minutes.

Inclusion criteria

* Children born in France aged 16 days to 24 months at the time of inclusion;
* Both parents born in a homogeneous geographical area: Sub-Saharan African countries;
* Children with no known pathology;
* Birth from 37 SA and before 42 SA;
* Birth weight greater than or equal to 2kg500 ;
* Apgar score at 10 to 5 minutes after birth;
* No opposition to data collection from holders of parental authority.

Non-inclusion criteria Not applicable

Study location Barthélemy Durand Hospital at Etampes, France

Results and Outcome Confirmation of the existence of specific psychomotor development characteristics in children born in France to parents born in Sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Children born in France, aged 16 days to 24 months at the time of inclusion
* Both parents born in a geographically homogeneous area: Sub-Saharan African countries
* Children with no known medical conditions
* Born between 37 and 42 weeks of gestational age
* Birth weight equal to or greater than 2.5 kg
* Apgar score of 10 at 5 minutes after birth
* No objection from the holders of parental authority to the collection of data

Exclusion Criteria:

* Not Applicable

Ages: 16 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children subjects from 16 days to 24 months, born in France to parents born in Sub-Saharan Africa
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Verify the existence of specific characteristics in the motor development of children born in France to parents born in Sub-Saharan Africa. | Between 60 and 90 minutes
  The primary outcome is to determine whether there are any specific characteristics exist in the motor development of children born in France to parents from Sub-Saharan Africa by comparing their average raw scores on the BSID-4 motor scale with the the French norms.

SECONDARY OUTCOMES:
Establish a developmental timeline for psychomotor skills in children born in France to parents born in Sub-Saharan Africa, based on 23 items from the early screening developmental norms provided by the government to early childhood professionals. | Between 60 and 90 minutes
  The development timeline for psychomotor skills in children born in France to parents born in Sub-Saharan Africa will be determined by calculating the average age of acquisition in the study's population for : Head control ; Grasps a presented object ; Social smile ; Reacts when spoken to ; Babbling ; Sitting unsupported ; Pulls to stand ; Moves independently (crawling, creeping, or other forms of movement) ; Imitation ; Independent walking ; Object permanence ; Thumb-index finger pincer grasp ; Turns head when name is called ; Reaction to the word "no" ; First word ; Joint attention ; Symbolic gestures ; Stacking blocks ; Points to a named object ; First phrases ; Proto-imperative pointing ; Running ; Kicking a ball.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Aguillon, Principal Investigator — Établissement Public de Santé Barthélemy Durand
Locations (1):
- Établissement Public de Santé Barthélemy Durand, Étampes, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cromwell EA, Dube Q, Cole SR, Chirambo C, Dow AE, Heyderman RS, Van Rie A. Validity of US norms for the Bayley Scales of Infant Development-III in Malawian children. Eur J Paediatr Neurol. 2014 Mar;18(2):223-30. doi: 10.1016/j.ejpn.2013.11.011. Epub 2013 Dec 31. PMID 24423629
- [Background] Rabain-Jamin J, Wornham WL. [Changes in maternal behavior and care practices in migrant women from Western Africa]. Psychiatr Enfant. 1990;33(1):287-319. French. PMID 2277816
- [Background] Karasik LB, Adolph KE, Tamis-Lemonda CS, Bornstein MH. WEIRD walking: cross-cultural research on motor development. Behav Brain Sci. 2010 Jun;33(2-3):95-6. doi: 10.1017/S0140525X10000117. Epub 2010 Jun 15. PMID 20546664
- [Background] Aina OF, Morakinyo O. Normative data on mental and motor development in Nigerian children. West Afr J Med. 2005 Apr-Jun;24(2):151-6. doi: 10.4314/wajm.v24i2.28187. PMID 16092318
- See also: Batista Wiese, E., Van Dijk, M., & Seddik, H. (2009). La matrice familiale dans l'immigration : trauma et résilience. Dialogue, 67-78. — https://shs.cairn.info/revue-dialogue-2009-3-page-67?lang=fr&ref=doi
- See also: Nguefack, S., Mbanga, V., & Mbassi, A. (2017). Développement psychomoteur d'une population de nourrissons camerounais à Yaoundé. Afrique Pédiatre génétique médicale, 26-33. — https://www.sobeped.com/wp-content/uploads/2024/02/4Developpement-psychomoteur-26-33.pdf